CLINICAL TRIAL: NCT03230071
Title: Efficacy and Safety of Twice Daily TMBCZG in Mild to Moderate Vascular Dementia: Randomized, Double Blind, Parallel Group, Placebo Controlled, Multicenter Trial
Brief Title: Efficacy and Safety of TMBCZG in Mild to Moderate Vascular Dementia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dongzhimen Hospital, Beijing (Other)
Collaborators: Beijing Union pharmaceutical factory II (Unknown); Beijing Compete Medical Technology Development Co. Ltd. (Unknown)
Responsible Party: Principal Investigator, Jinzhou Tian, vice-president, Dongzhimen Hospital, Beijing
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P2017-03-BDY-03-V03
Record Dates: First submitted 2017-07-24; First posted 2017-07-26 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-02

CONDITIONS: Vascular Dementia
Keywords: Herbal therapy; Randomized controlled trial; Vascular Dementia
MeSH Terms: conditions — Dementia, Vascular

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): placebo identified to TMBCZG,0.1g per pill which contains 0mg TMBCZG，3 pills per time, 2 times per day for 24 weeks.
  Interventions: Other: placebo
- TMBCZG-high dose (Experimental): TMBCZG, 0.1g per pill which contains 14mg TMBCZG, 3 pills per time, 2 times per day for 24 weeks.
  Interventions: Drug: TMBCZG
- TMBCZG-medium dose (Experimental): TMBCZG( 0.1g per pill which contains 14mg TMBCZG) and placebo identified to TMBCZG(0.1g per pill which contains 0mg TMBCZG), 2 TMBCZG pills and 1 placebo pill per time, 2 times per day for 24 weeks.
  Interventions: Drug: TMBCZG; Other: placebo
- TMBCZG-low dose (Experimental): TMBCZG( 0.1g per pill which contains 14mg TMBCZG) and placebo identified to TMBCZG(0.1g per pill which contains 0mg TMBCZG), 1 TMBCZG pills and 2 placebo pill per time, 2 times per day for 24 weeks.
  Interventions: Drug: TMBCZG; Other: placebo

INTERVENTIONS:
Drug: TMBCZG — 0.1g per pill which contains 14mg TMBCZG
  Other Names: TianMaBianChunZhiGanPian; TianMaYouJiDuoSuanBianZhiGanPian(TMYJDSBZG)
  Arms: TMBCZG-high dose; TMBCZG-low dose; TMBCZG-medium dose
Other: placebo — 0.1g per pill which contains 0mg TMBCZG
  Arms: Placebo; TMBCZG-low dose; TMBCZG-medium dose

SUMMARY:
The study will be a 24-week multicentre, double-blind, placebo-controlled phase Ⅱa trial with 4 treatment arms in China. Participants aged 55-80 years will be randomized to TMBCZG-high dose(84mg per day), TMBCZG- medium dose(56mg per day), TMBCZG- low dose(28mg per day) or to placebo. The primary endpoint will be VADAS-Cog and CDR-SB. Secondary outcomes included changes in MMSE and ADL. Patients' safety will be assessed by recording of adverse events, clinical examinations, electrocardiography and laboratory tests. The patients, caregivers, and investigators will be blinded to the treatment allocations.

ELIGIBILITY:
Inclusion Criteria:

* Patients meeting the clinical diagnosis of probable vascular dementia(VaD) established according to the National Institute of Neurological Disorders and Stroke and the Association Internationale pour la Recherche et l'Enseignement en Neurosciences (NINDS-AIREN)were eligible to participate:

  1. Dementia defined by clinical core criteria,
  2. Cerebrovascular disease, defined by history of stroke, as well as multiple basal ganglia and white matter lacunes, or extensive periventricular white matter lesions( excluded medial temporal lobe atrophy or other special image),
  3. A relationship between dementia and Cerebrovascular disease, manifested or inferred by the presence of one or more of the following: (a) onset of dementia within 3 months following a recognized stroke; (b) abrupt deterioration in cognitive functions; or fluctuating, stepwise progression of cognitive deficits.
* Mild to Moderate Dementia with MMSE score of ≤26 and ≥11;
* Aged ≥55 and ≤80 years old in both gender;
* Weighing of ≥45kg and ≤90kg;
* Adequate vision and hearing ability to complete all study tests;
* With a stable caregiver.
* Have a certain level of language competence (can read simple articles and write simple sentences);
* Informed consent, signed informed consent by legal guardian.

Exclusion Criteria:

* A medical history of other dementia types, like mixed dementia, Alzheimer's disease, frontotemporal dementia, Parkinson's disease dementia, dementia with Lewy bodies, Huntington disease, et al;
* Subdural hematoma, traffic hydrocephalus, brain tumor, thyroid disease,vitamin deficiency or other diseases which can lead to cognitive impediment;
* Major depression (HAMD≥17) or major anxious(HAMA≥12);
* Subject can't complete related test due to severe neurologic deficits, such as hemiplegia, aphasia, audio-visual disorder and so forth;
* Severe cardiovascular disease(severe arrhythmia, myocardial infarction within 3 months, New York Heart Association Functional Classification III-IV, systolic pressure≥180mmHg or ≤90mmHg);
* Severe liver or kidney dysfunction (alanine aminotransferase or aspartate transaminase is more than 1.5 times the upper limit of normal, or serum creatinine is more than the upper limit of normal);
* Uncontrolled diabetes(glycosylated hemoglobin is more than 2 times the upper limit of normal);
* Asthma, chronic obstructive pulmonary disease, multiple neuritis, myasthenia gravis and muscle atrophy;
* Severe indigestion, gastrointestinal obstruction, gastric and duodenal ulcers and other gastrointestinal disorders that can affect drug absorption;
* A medical history of epileptic history, glaucoma, alcoholism, or psycho-substance abuse;
* Subject has been taking cholinesterase inhibitors, memantine, nimodipine or herbal medicine with function of improving cognition in the past one month;
* Use of sympathomimetic or antihistamines drugs within 48h before assessment;
* Allergic constitution or allergic reactions to experimental drug;
* According to the assessment of the investigator, subject cann't complete the study due to poor compliance or other reasons;
* Subject is participating in other clinical trials or participated in the past 1 month.

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2017-07-28 (Actual); Primary Completion 2019-08-22 (Actual); Study Completion 2021-02-05 (Actual)

PRIMARY OUTCOMES:
Vascular Dementia Assessment Scale-cognitive subscale(VADAS-Cog) | baseline, 4-week, 12-week, 24-week and 28-week.
  Change from baseline to end of double-blind treatment of VADAS-Cog.
Clinical Dementia Rating-Sum of Boxes (CDR-SB) | baseline, 4-week, 12-week, 24-week and 28-week.
  Change from baseline to end of double-blind treatment of CDR-SB.

SECONDARY OUTCOMES:
Mini-Mental State Examination (MMSE) | baseline, 4-week, 12-week, 24-week and 28-week.
  Change from baseline to end of double-blind treatment of MMSE.
Activities of daily living (ADL) | baseline, 4-week, 12-week, 24-week and 28-week.
  Change from baseline to end of double-blind treatment of ADL.

CONTACTS AND LOCATIONS:
Overall Officials: JinZhou Tian, MD,PhD, Study Director — Dongzhimen Hospital, Beijing
Locations (1):
- Dongzhimen Hospital ,Beijing University of Chinese Medicine, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tian J, Shi J, Wei M, Li T, Ni J, Zhang X, Zhang M, Li Y, Wang Y. Efficacy and safety of Tianmabianchunzhigan in mild to moderate vascular dementia: Protocol of a randomized controlled IIa trial. Medicine (Baltimore). 2018 Dec;97(51):e13760. doi: 10.1097/MD.0000000000013760. PMID 30572524